CLINICAL TRIAL: NCT01791933
Title: The Evaluation of the Effectiveness of CAM Treatments for Lumbar and Cervical Spine Pain Patients Due to Spinal Disease : Prospective, Observational Study
Brief Title: The Evaluation of the Effectiveness of CAM Treatments for Lumbar and Cervical Spine Pain Patients Due to Spinal Disease
Status: Completed | Type: Observational
Sponsor: Jaseng Hospital of Korean Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2013-01
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Lumbar and Cervical Pain
Keywords: LBP; Neck pain; Integrative package; CAM
MeSH Terms: conditions — Neck Pain | interventions — Phytotherapy; Acupuncture Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CAM treatment
  Interventions: Drug: herbal medicine; Procedure: Chuna manual therapy; Procedure: Acupuncture; Procedure: Bee-venom pharmacoacupuncture/pharmacoacupuncture

INTERVENTIONS:
Drug: herbal medicine — 120ml of Chuna herbal medicine(Ostericum koreanum, Eucommia ulmoides, Acanthopanax Sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, and Cuscuta chinensis) taken twice a day 30 minutes after meals for more than 2 months
Procedure: Chuna manual therapy — A type of Korean spinal manual therapy administered 5~10 minutes at physician's discretion 1-2times a week for more than 2 months Applies mobilization using High-Velocity, Low-Amplitude thrusts to joints slightly beyond the passive ROM and manual force within the passive ROM without thrusts.
  Other Names: Chuna manipulation
Procedure: Acupuncture — Acupuncture using sterilized disposable needles, sized 0.30X40mm. Needles left for 15~20 minutes, selecting 6 acupoints(both BL23, BL24, BL25 ) and other acupoints at physician's discretion, using a total of 10~20 acupoints 1-2times a week for more than 2 months
Procedure: Bee-venom pharmacoacupuncture/pharmacoacupuncture — pharmacoacupuncture using 30G sterilized bee venom. Selecting 6 acupoints(both BL23, BL24, BL25) and other acupoints at physician's discretion, concentration 10,000:1, 0.1 cc per acupoint, total amount injected 1.0 cc/session 1-2times a week for more than 2 months
  Other Names: BV; Bee-venom therapy

SUMMARY:
The purpose of this study is to investigate the effect of CAM treatments consisting of herbal medicine, Chuna manual therapy, pharmacoacupuncture, acupuncture on lumbar and cervical spine pain patients due to spinal disease.

DETAILED DESCRIPTION:
"The purpose of this study is to investigate the effect of CAM treatments on lumbar and cervical spine pain patients due to spinal disease.

After subjects selected by screening, who receive CAM treatments 1-2times a week for more than 2 months and F/U at 1st, 2nd, 3rd month by meeting and F/U at 6nd, 12nd month by calling.

The CAM treatments used in this study consists of 120ml of Chuna herbal medicine(Ostericum koreanum, Eucommia ulmoides, Acanthopanax Sessiliflorus, Achyranthes bidentata, Psoralea corylifolia, Peucedanum japonicum, Cibotium barometz, Lycium chinense, Boschniakia rossica, and Cuscuta chinensis) and dried extracts in pill form(Cibotium barometz, Atractylodes japonica) taken twice a day 30 minutes after meals, Chuna manual therapy, intermuscular injections of bee-venom pharmacoacupuncture(Select 6 acupoints, concentration 10,000:1, 0.1 cc per acupoint, total amount injected 1.0 cc/session), acupuncture and allow for NSAID intake during the investigational period. The subject is allowed a maximum of 3 pills/day, taken at a minimum of 8 hrs apart. The number of pills taken will be measured at 4 wks after conclusion of treatment."

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from low back pain or Neck due to spinal disease Agree to the treatment of more than 2 months
* Age all(If under 18yr, Guardian's consent need)
* Volunteers do not have a problem with my speech as those who have signed the consent

Exclusion Criteria:

* Diagnosis of serious disease(s) which are possible causes of back pain such as malignancy, vertebral fracture, spinal infection, inflammatory spondylitis, cauda equina compression, etc.
* Prior diagnosis of other chronic disease(s) which could affect effectiveness or interpretation of treatment results such as cardiovascular disease, diabetic neuropathy, fibromyalgia, rheumatoid arthritis, Alzheimer's disease, epilepsy, etc.
* Progressive neurologic deficit(s) or concurrent severe neurological symptoms Unsuitable for or at risk of complications from acupuncture treatment such as patients with clotting disorders, severe diabetes with risk of infection, serious cardiovascular disease, or undergoing anticoagulant treatment, etc.
* Under prescription of corticosteroids, immuno-suppressant drugs, psychiatric medicine, or other medication considered unsuitable for subjects by the researcher
* Experience of gastroenteric complications after taking NSAIDs or currently undergoing treatment for digestive disorders
* During pregnancy or suspected pregnancy
* Subjects considered unsuitable for clinical trial by the researcher

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patient sampling within lumbar and cervical spine pain patients due to spinal disease.
Sampling Method: Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
NRS of low back pain or neck pain/NRS of radiating pain | Change from Baseline at 3rd month

SECONDARY OUTCOMES:
ODI (Oswestry Disability Index) | Baseline, 1st month, 2nd month, 3rd month
Patient satisfaction | 3rd month
  Patient satisfaction of treatment
Job loss | Baseline, 1st month, 2nd month, 3rd month
  Life activity of loss rate
painkiller intaken of times | Baseline, 3rd month
Adverse reactions | Baseline, 1st month, 2nd month, 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Jinho LEE, KMD, Principal Investigator — Jaseng Hospital of Korean Medicine
Locations (1):
- Jaseng Hospital of Oriental Medicine, Seoul, Gangnam-gu, South Korea